CLINICAL TRIAL: NCT04200001
Title: Evaluation of Sexual Quality of Life in Women Less Than 51 Years Old, During Adjuvant Hormonal Therapy for Breast Cancer
Brief Title: Evaluation of Sexual Quality of Life for Breast Cancer
Acronym: CUPIDON2
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2019-16-BCU
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Cancer; Quality of Life
Keywords: breast cancer; hormonotherapy; women; quality of life
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adjuvant hormonal therapy for breast cancer: women less than 51 years old, during adjuvant hormonal therapy for breast cancer
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — The patient will receive the following questionnaires to be completed :
  * EORTC QLQ-C30
  * EORTC QLQ-BR23
  * EORTC SHQ-C22
  * CUPIDON 2 specific questionnaire

SUMMARY:
Breast cancer is the most common cancer in women worldwide. Hormonal therapy is one of the major treatments for hormone receptor positive breast tumors. It is prescribed to 70% of breast cancer patients. Hormonal therapy can be responsible for sexual dysfunction induced by hormonal changes. Extended adjuvant hormonal therapy over 5 years increases these adverse effects.

According to the third "Plan Cancer" (2014-2019), sexual dysfunction prevention and screening must be systematic as an integral part of supportive care. Nevertheless, sexual quality of life remains too rarely considered.

In this study, the investigator propose to evaluate sexual quality of life of women less than 51 years old during the adjuvant endocrine therapy for localized breast cancer. The investigator also intend to collect the supportive measures or interventions used by women to overcome sexual dysfunction. Finally, this study aims to evaluate the need for sexual trouble specific management and acceptability of different methods.

This project is a hot topic as the interest for oncosexuality is growing, and the need for specific management is increasing with still insufficient access to specific care.

DETAILED DESCRIPTION:
In 2006, the World Health Organization provided a definition of sexual health stating that "for sexual health to be reached and maintained, the sexual rights of all persons must be respected and fulfilled". Sexual quality of life is now an admitted and relevant parameter of global health and global quality of life.

The VICAN 2 (Vie après le CANcer 2 years after diagnosis) survey showed that 2/3 of the sexually active French breast cancer survivors reported impaired sexual health, persisting 2 years after cancer diagnosis.

The deterioration of sexual health is multifactorial: (1) psychological: body image, sexual identity; (2) physiological: sexual functionality, steps of the feminine sexual response; (3) familial, social and professional. The alteration of sexuality is mainly due to cancer treatments: surgery, radiotherapy, chemotherapy and endocrine therapy.

Breast cancer is the most common cancer in women worldwide. Hormonal therapy is one of the major treatments for hormone receptor positive breast tumors. It is prescribed to 70% of breast cancer patients. Hormonal therapy can be responsible for sexual dysfunction induced by hormonal changes. Extended adjuvant hormonal therapy over 5 years increases these adverse effects.

According to the third "Plan Cancer" (2014-2019), sexual dysfunction prevention and screening must be systematic as an integral part of supportive care. Nevertheless, sexual quality of life remains too rarely considered.

In this study, the investigator propose to evaluate sexual quality of life of women less than 51 years old during the adjuvant endocrine therapy for localized breast cancer. The investigator also intend to collect the supportive measures or interventions used by women to overcome sexual dysfunction. Finally, this study aims to evaluate the need for sexual trouble specific management and acceptability of different methods.

This project is a hot topic as the interest for oncosexuality is growing, and the need for specific management is increasing with still insufficient access to specific care.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥ 18 years old and less than 51 years old.
* Patient with non-metastatic early breast cancer,
* Patient undergoing adjuvant hormonal therapy for at least 2 years,
* Patient who has been treated by surgery, with or without chemotherapy and/or radiotherapy.
* Patient being currently sexually active.
* Patient who agreed, after receiving information, to participate to the study.

Exclusion Criteria:

* Patient who refused to participate to this study or is unable to fulfill a questionnaire,
* Patient not affiliated to the French social security system,
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation,
* Patient whose regular monitoring is impossible for psychological, family, social or geographical reasons,
* Pregnant and / or breastfeeding woman.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women less than 51 years old, during adjuvant hormonal therapy for breast cancer.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Sexual quality of life: EORTC SHQ-C22 questionnaire | At the inclusion, at one time
  Sexual quality of life assessed by the EORTC SHQ-C22 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Véronique D'HONDT, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pouget JP, Lozza C, Deshayes E, Boudousq V, Navarro-Teulon I. Introduction to radiobiology of targeted radionuclide therapy. Front Med (Lausanne). 2015 Mar 17;2:12. doi: 10.3389/fmed.2015.00012. eCollection 2015. PMID 25853132
- [Background] Kumar C, Shetake N, Desai S, Kumar A, Samuel G, Pandey BN. Relevance of radiobiological concepts in radionuclide therapy of cancer. Int J Radiat Biol. 2016;92(4):173-86. doi: 10.3109/09553002.2016.1144944. Epub 2016 Feb 26. PMID 26917443